CLINICAL TRIAL: NCT01122277
Title: Klinisches Register RaFTinG - Rational Fluid Therapy in Germany
Brief Title: Rational Fluid Therapy in Germany
Acronym: RaFTinG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: University Hospital Muenster (Other); Fresenius Kabi, Bad Homburg, Germany (Unknown)
Responsible Party: PD Dr. Matthias Jacob, Klinikum der Universität München, Klinik für Anaesthesiologie
Other Study IDs: 337 -09/2009-366-f-S
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2010-10

CONDITIONS: Patients in ICU
Keywords: Volume therapy; Fluid therapy; Patients in ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is the prospective documentation and evaluation of the status quo of volume therapy in German intensive care units.

DETAILED DESCRIPTION:
The purpose of RaFTinG is the prospective documentation and evaluation of the demographic, diagnostic and therapeutic characteristics of unselected patients and their treatment in intensive care units (ICU) in Germany.

Documentation will not only include their stay in the ICU but a follow up query 90 days after discharge from the ICU.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with an indication for fluid/volume therapy

Exclusion Criteria:

* Patients hospitalized by order of a court of law or a government agency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care units with an indication for fluid/volume therapy
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Jacob, MD, Principal Investigator — Klinik für Anaesthesiologie, Klinikum der Universität München; Christian Ertmer, MD, Principal Investigator — Universitätsklinikum Münster, Germany; Bernhard Zwissler, Prof, Study Chair — Klinik für Anaesthesiologie, Klinikum der Universität München, Germany; Hugo van Aken, Prof, Study Chair — Universitätsklinikum Münster, Germany
Locations (2):
- Germany (2):
  - Klinik für Anaesthesiologie, Klinikum der Universität München, Munich, Bavaria
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia

REFERENCES:
- [Derived] Ertmer C, Zwissler B, Van Aken H, Christ M, Spohr F, Schneider A, Deisz R, Jacob M. Fluid therapy and outcome: a prospective observational study in 65 German intensive care units between 2010 and 2011. Ann Intensive Care. 2018 Feb 17;8(1):27. doi: 10.1186/s13613-018-0364-z. PMID 29455308